CLINICAL TRIAL: NCT00763672
Title: Impact of a Single Second-trimester Plasma sFlt-1 and/or Urinary PlGF Assay on Maternofetal Morbidity/Mortality
Brief Title: MorbiMortality Amelioration in Preeclamptic Primiparas Study. MoMA Pre Prim Study
Acronym: MOMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P051060
Record Dates: First submitted 2008-09-30; First posted 2008-10-01 (Estimated); Last update posted 2013-03-28 (Estimated); Status verified 2013-03

CONDITIONS: Pregnancy; Primiparity; Hypertension; Preeclampsia; Intrauterine Growth Retardation
Keywords: Preeclampsia; Hypertension; Intra uterine growth retardation; Antiangiogenic factor; Prevention
MeSH Terms: conditions — Hypertension; Pre-Eclampsia; Fetal Growth Retardation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Other): sFlt-1 status known
  Interventions: Other: Transmission of sFlt-1 results to the investigator
- B (Other): sFlt-1 status unknown
  Interventions: Other: No transmission of the sFlt-1 results to the investigator

INTERVENTIONS:
Other: Transmission of sFlt-1 results to the investigator — Transmission of sFlt-1 results by the laboratory to the investigator
  Other Names: Transmission of sFlt-1
  Arms: A
Other: No transmission of the sFlt-1 results to the investigator — The laboratory do not transmit the sFlt-1 results to the investigator before the end of the study.
  Other Names: No transmission of the sFlt-1
  Arms: B

SUMMARY:
The purpose of this study is to determine whether close monitoring of patients with a high sFlt1 plasma level between 25 and 28 weeks of gestation (i.e. at high risk of subsequent preeclampsia) improves maternal and fetal outcomes. The investigator hypothesize that 1/ early screening for preeclampsia by plasmatic sFlt1 will reduce maternal and fetal mortality and morbidity and 2/ a simple urinary PlGF screening will be effective.

DETAILED DESCRIPTION:
We will measure plasmatic sFlt-1 level between 25 and 28 weeks of gestation and flow velocity of uterine arteries by Doppler (22 - 26 weeks of gestation) in primipara. Patients will be stratified according to the results of the uterine artery Doppler measurement, and then randomized in two groups A and B. In group A, sFlt-1 concentration will be communicated to the obstetrician (+ or -): the threshold of abnormally high plasmatic concentration of sFlt-1 is 957 ng/mL. In patients with a high plasmatic concentration of sFlt-1 (+), the pregnancy will be closely monitored including repeated clinical, biological, and ultrasound examinations. Patients with sFlt-1 plasmatic concentration below 957 ng/mL (-) will be routinely followed-up.In group B, the result of sFlt-1 measurement will not be communicated and the pregnancy will be routinely monitored.Abnormal Doppler recordings in either group will result in a close monitoring as per our usual local practice. Urinary PlGF (expressed as a ratio PlGF/creatininemia) will also be measured and the results will be analyzed at the end of the study. Beside sFlt-1, we will store the plasmatic samples to measure other biomarkers that could be relevant in the future (no DNA analysis will be done without a new patient consent).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant womenAge ≥ 18 years
* Followed in our center before the 28th week of gestation
* Under social security coverage
* Signed informed consent

Exclusion Criteria:

* Age < 18 years
* Followed in our center after the 28th week of gestation
* No social security coverage
* Refusal to be included

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1040 (Actual)
Dates: Start 2008-11; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Reduction in the maternal and fetal morbimortality score | During the pregnancy and the 3 first month of the child

SECONDARY OUTCOMES:
Child status | at 3 months post-delivery
Length of hospital stay during pregnancy and post-partum periods | during pregnancy and post-partum periods
Predictive value for vascula-renal disease of urinary PlGF as compared with plasmatic sFlt-1. | between 25 and 28 weeks of gestation

CONTACTS AND LOCATIONS:
Overall Officials: Nadia BERKANE, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Department of Gynecology Obstetrics and Reproductive Medicine, Hôpital Tenon, AP-HP, UPMC, Paris, France

REFERENCES:
- [Background] Sibai B, Dekker G, Kupferminc M. Pre-eclampsia. Lancet. 2005 Feb 26-Mar 4;365(9461):785-99. doi: 10.1016/S0140-6736(05)17987-2. PMID 15733721
- [Background] Nagamatsu T, Fujii T, Kusumi M, Zou L, Yamashita T, Osuga Y, Momoeda M, Kozuma S, Taketani Y. Cytotrophoblasts up-regulate soluble fms-like tyrosine kinase-1 expression under reduced oxygen: an implication for the placental vascular development and the pathophysiology of preeclampsia. Endocrinology. 2004 Nov;145(11):4838-45. doi: 10.1210/en.2004-0533. Epub 2004 Jul 29. PMID 15284201
- [Background] Familoni OB, Adefuye PO, Olunuga TO. Pattern and factors affecting the outcome of pregnancy in hypertensive patients. J Natl Med Assoc. 2004 Dec;96(12):1626-31. PMID 15622693
- [Background] Maynard SE, Min JY, Merchan J, Lim KH, Li J, Mondal S, Libermann TA, Morgan JP, Sellke FW, Stillman IE, Epstein FH, Sukhatme VP, Karumanchi SA. Excess placental soluble fms-like tyrosine kinase 1 (sFlt1) may contribute to endothelial dysfunction, hypertension, and proteinuria in preeclampsia. J Clin Invest. 2003 Mar;111(5):649-58. doi: 10.1172/JCI17189. PMID 12618519
- [Background] Sugimoto H, Hamano Y, Charytan D, Cosgrove D, Kieran M, Sudhakar A, Kalluri R. Neutralization of circulating vascular endothelial growth factor (VEGF) by anti-VEGF antibodies and soluble VEGF receptor 1 (sFlt-1) induces proteinuria. J Biol Chem. 2003 Apr 11;278(15):12605-8. doi: 10.1074/jbc.C300012200. Epub 2003 Jan 21. PMID 12538598
- [Background] Luttun A, Carmeliet P. Soluble VEGF receptor Flt1: the elusive preeclampsia factor discovered? J Clin Invest. 2003 Mar;111(5):600-2. doi: 10.1172/JCI18015. No abstract available. PMID 12618513
- [Background] Koga K, Osuga Y, Yoshino O, Hirota Y, Ruimeng X, Hirata T, Takeda S, Yano T, Tsutsumi O, Taketani Y. Elevated serum soluble vascular endothelial growth factor receptor 1 (sVEGFR-1) levels in women with preeclampsia. J Clin Endocrinol Metab. 2003 May;88(5):2348-51. doi: 10.1210/jc.2002-021942. PMID 12727995
- [Background] Romero R, Nien JK, Espinoza J, Todem D, Fu W, Chung H, Kusanovic JP, Gotsch F, Erez O, Mazaki-Tovi S, Gomez R, Edwin S, Chaiworapongsa T, Levine RJ, Karumanchi SA. A longitudinal study of angiogenic (placental growth factor) and anti-angiogenic (soluble endoglin and soluble vascular endothelial growth factor receptor-1) factors in normal pregnancy and patients destined to develop preeclampsia and deliver a small for gestational age neonate. J Matern Fetal Neonatal Med. 2008 Jan;21(1):9-23. doi: 10.1080/14767050701830480. PMID 18175241
- [Background] Stepan H, Geide A, Faber R. Soluble fms-like tyrosine kinase 1. N Engl J Med. 2004 Nov 18;351(21):2241-2. doi: 10.1056/NEJM200411183512123. No abstract available. PMID 15548791
- [Background] Levine RJ, Maynard SE, Qian C, Lim KH, England LJ, Yu KF, Schisterman EF, Thadhani R, Sachs BP, Epstein FH, Sibai BM, Sukhatme VP, Karumanchi SA. Circulating angiogenic factors and the risk of preeclampsia. N Engl J Med. 2004 Feb 12;350(7):672-83. doi: 10.1056/NEJMoa031884. Epub 2004 Feb 5. PMID 14764923
- [Background] Hertig A, Berkane N, Lefevre G, Toumi K, Marti HP, Capeau J, Uzan S, Rondeau E. Maternal serum sFlt1 concentration is an early and reliable predictive marker of preeclampsia. Clin Chem. 2004 Sep;50(9):1702-3. doi: 10.1373/clinchem.2004.036715. No abstract available. PMID 15331514
- [Background] Levine RJ, Thadhani R, Qian C, Lam C, Lim KH, Yu KF, Blink AL, Sachs BP, Epstein FH, Sibai BM, Sukhatme VP, Karumanchi SA. Urinary placental growth factor and risk of preeclampsia. JAMA. 2005 Jan 5;293(1):77-85. doi: 10.1001/jama.293.1.77. PMID 15632339
- [Background] Berkane N, Hertig A, Rondeau E, Uzan S. Hypertensive disorders of pregnancy: future perspectives. A French point of view. Curr Opin Obstet Gynecol. 2008 Apr;20(2):107-9. doi: 10.1097/GCO.0b013e3282f73391. No abstract available. PMID 18388807